CLINICAL TRIAL: NCT06923865
Title: Now! Project - a Controlled Evaluation of a Physical Activity Program for Adolescents With Overweight
Brief Title: Controlled Evaluation of an Exercise Program for Overweight Adolescents
Acronym: Now!
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Gesundheitsförderung Schweiz, GFCH (Unknown); University of Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Now!-Projekt, 2024-01651
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Adolescent; Pediatric Obesity; Exercise Therapy; Health Promotion; Program Evaluation; Impulse Control Disorders; Quality of Life; Retinal Vessels; Strength Training Effects; Aerobic Capacity
Keywords: Overweight adolescents; Youth physical activity; Motor performance in children; Impulse control and fitness; training in peer groups
MeSH Terms: conditions — Pediatric Obesity; Disruptive, Impulse Control, and Conduct Disorders | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Active Comparator): training group: Two peer-group sessions per week, each including at least 90 minutes of training/workout involving moderate to vigorous physical activity.
  Interventions: Behavioral: training group
- control group (No Intervention): There is no intervention in the control group. The control group only receives the WHO physical activity recommendations as well as the results of the assessments in the form of a detailed health report.
  Control arm: Observation of physical and psychological development without additional intervention.

INTERVENTIONS:
Behavioral: training group — Participants in training group are invited to take part in two structured training sessions per week, each lasting 90 minutes:
  One session takes place in a larger group setting, where participants engage in physical activities and games together.
  The second session is held in a small group format with 1-2 peers-either friends the participant already knows or peers they meet during the larger group session.
  Each training session is supervised by a qualified instructor and includes:
  Fun, game-based activities
  Short workouts aimed at improving fitness
  A focus on social interaction, enjoyment, and participation
  The sessions are designed to be supportive, engaging, and motivating, with the goal of increasing physical activity in a positive group environment.
  Arms: training group

SUMMARY:
Physical activity decreases as young people get older, especially during the shift from early to late adolescence. Unfortunately, around 81% of school-aged children worldwide between the ages of 11 and 17 do not meet the recommendation of at least one hour of physical activity per day - and this is also true in Switzerland. Not being active enough, whether normal weight or overweight, can lead to long-term health problems and is a major factor in becoming overweight over time. This results in healthcare costs and negatively affects quality of life. Supporting physical activity in overweight youth requires well-rounded, thoughtful programs.

The investigators studying the impact of the movement programs now! and now!+ on the physical activity and health of young people. The goal is to look at both physical and mental changes equally.

Taking part in this study involves minimal physical or mental risk for the participants. These small risks from the testing methods and activities are taken into account in how the program is explained and carried out.

The benefits for the participants - feeling healthier and fitter physically, and more confident and capable mentally - clearly outweigh any potential risks, thanks to the additional, guided, and personalized exercise program.

The participants take part in the now! and now!+ exercise programs run by the Basel-Stadt Sports Office and the DSBG. now! is a 90-minute group session with up to 14 young people, while now!+ is a 90-minute small-group session with 2 to 4 participants. Both programs take place once a week over a 12-month period and pause during school holidays (38 training weeks in total).

Each session includes a warm-up, a strength or endurance training block, and a coordination phase. The program is modular and adapted to the physical and personal needs of each participant. This ensures that overweight adolescents are not overstrained and don't develop symptoms like pain, frustration, or lack of motivation (Behringer et al., 2011), while still allowing for a training stimulus that supports physical improvement.

The results of the evaluations are directly used to improve and further develop the exercise program. The overall project includes three rounds, each consisting of one year of training and three test sessions, each lasting about two hours. The now! and now!+ programs are held weekly for a total of 38 weeks per year, with breaks during school holidays.

Each of the three test sessions includes the same set of assessments (see "Study Intervention") and follows a set order: The process begins with measuring body size and blood pressure, followed by a static retinal vessel analysis. After these medical checks, participants do a 5-minute warm-up on a stationary bike at a set resistance level. Then, strength tests are performed: knee extension on the IsoMed 2000, handgrip strength, and jump power on the Leonardo force plate. The endurance test using spiroergometry marks the end of the physical assessments.

Finally, impulse control is tested, and participants complete a set of questionnaires. At the end of the session, each participant is given an actigraph (a small motion sensor worn on the body) to track their physical activity over the following seven days.

ELIGIBILITY:
Inclusion Criteria:

* BMI above the 90th percentile for their age and gender (WHO reference table)
* Deficits in movement motivation and motor skills
* No health complaints or movement-restricting conditions
* No health risks for maximal exertion
* Ability to verbally communicate pain or discomfort
* Unremarkable PAR-Q questionnaire
* Signed parental consent form

Exclusion Criteria:

* Acute or chronic illness
* Inability to follow the study procedures (e.g., language barriers, psychological disorders)

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Aerobic performance | over the time period of one year of intervention, october to october
  Cardiopulmonary exercise testing (CPET) will be performed on a mechanically braked bicycle ergometer (Ergoselect 200, Ergoline GmbH, Germany). Ventilation and gas exchange will be measured breath-by-breath using a face mask connected to a Cortex Metalyzer 3B (Cortex Biophysik GmbH, Germany). Basic spirometry is conducted before testing. A 12-lead ECG (Customed GmbH, Germany) is used at rest and during exercise to monitor heart rate and detect abnormalities. CPET begins with a 3-minute resting phase and continues using one of five established protocols (Wagner et al., 2019). Participants are verbally encouraged throughout. Gas exchange values are averaged every 30 seconds. VO₂max and RERmax are recorded as peak values at or before exhaustion. Subjective exertion is assessed every 2 minutes and post-exercise using the Borg scale (Borg, 1998).
Strength assessment | over the time period of one year of intervention, october to october
  The measurement of isometric maximal voluntary contraction of lower extremity muscles will be performed in a seated position in a dynamometer (Isomed 2000, D. & R. Ferstl GmbH, Hemau, Germany). This test is similar to a typical leg press commonly found in gyms. According to Maffiuletti et al. (2016) the subjects are instructed to extend their legs as fast and forceful as possible and hold the contraction for 3-5s. After a familiarization attempt, the measurement is performed three times with a rest of 45 s in between. Peak torque will be used as primary outcome.

SECONDARY OUTCOMES:
Retinal vessel Analysis | time period of one year
  Static retinal vessel diameters will be analysed using a Static Retinal Vessel Analyzer (SVA-T, IMEDOS Health GmbH, Jena, Germany). The system consists of a fundus camera (Topcon TRC NW8) and analysing software (Visualis, IMEDOS Health GmbH), allowing non-invasive and non-mydriatic assessment of retinal vessel diameters. Two valid images from the retina of the left and right eye with an angle of 45° and with the optic disc in the centre will be taken. Reti-nal arterioles and venules, coursing through an area of 0.5-1 disc diameter (d) from the optic disc margin, will be identified semi-automatically at higher magnification using special analysing software (Vesselmap 2, Visualis IMEDOS Health GmbH). Diameters will be averaged to central retinal arteriolar (CRAE) and venular (CRVE) diameters, using the Parr-Hubbard formula de-scribed elsewhere (Ikram et al., 2006) and the AVR will be calculated from the CRAE and CRVE. Retinal vessel diameters are generally presented in measuring units (
Blood pressure | time period of one year
  Blood pressure will be assessed in a supine position after a rest period of five minutes by use of a validated automated oscillograph (Mindray VS-900, Mindray, Darmstadt, Germany) for use in children and adolescents (Wong et al., 2006) Cuff size will be selected based on the individual circumference of the upper right arm according to the guidelines (Flynn et al., 2017; NHBPE Program, 2004). Blood pressure is measured 3 times with 2 min apart, whereby the last two are averaged and the first is discarded.
Enjoyment of physical activity | over the time period of one year of intervention, october to october
  To measure psychological acceptance, participants are asked to complete the Acceptance and Fusion Questionnaire for Youth (AFQ-Y). This instrument assesses the willingness to experience private events, values-oriented action, experiential avoidance, and cognitive and emotional fu-sion. The Difficulties in Emotion Regulation Scale (DERS-36) is used to measure difficulties in emotion regulation. Additional information on sleep behavior, perceived stress, and well-being is gathered using the Insomnia Severity Index (ISI), the Perceived Stress Scale-Youth (PSS-Y), and the WHO-5 Well-Being Index.
Body composition | over the time period of one year of intervention, october to october
  Body weight and composition in light clothing will be conducted using the gold-standard method, dual-energy x-ray absorptiometry (DEXA), utilizing a GE Lunar iDXA® device (GE Lunar Inc., Madison, WI; software version 13.10). Participants in the study are required to fast for 6 hours prior to the assessment. The analysis will yield both absolute and relative metrics for total body fat mass and fat-free mass. Throughout the assessment, subjects will lie in a supine position (Marra et al., 2019). The effective radiation dose from a single whole-body DEXA (<10 μSv) is similar to the normal background radiation received over one day at sea level.(Shepherd et al., 2017)

OTHER OUTCOMES:
Power assessment | over the time period of one year of intervention, october to october
  Power per body mass, determined from a vertical countermovement jump (CMJ), has been shown to be correlated to leg extension strength in children while representing a more natural movement. The CMJ will be performed on a force plate (Leonardo Mechanograph®, Novo-tec medical, Pforzheim, Germany) with arms akimbo. The instruction will be to jump as high as possible. After familiarization, each participant performs 5 trials, with the best of the two trials with <5% difference being used for the analysis. The most important outcome parameter of this test is the maximum power output (peak power) normalized to body weight. The CMJ had a high intra-trial reproducibility (ICC>0.95) in children, whereas inter-session variation has been re-ported to be high in prebubertal and early pubertal children as well (ICC=0.95, SEE=1.92 stand-ard error of estimate).
Handgrip Strength | over the time period of one year of intervention, october to october
  The handgrip strength is measured with an adjustable application to accommodate the span of each hand size (Leonardo Mechanograph®, Novotec medical, Pforzheim, Germany). The measurement is performed with the arm held vertically straight, providing a safe and reliable measurement for children (Gąsior et al., 2020). The subjects are instructed to compress the ad-justable application as forceful as possible and hold the contraction for 5s. After a familiarization attempt, the measurement is performed three times with a rest of 1 min in between.
Acceptance and Fusion Questionnaire for Youth (AFQ-Y) | over the time period of one year of intervention, october to october
  This self-report questionnaire assesses psychological acceptance in children and adolescents. It measures key components such as willingness to experience uncomfortable thoughts and emotions (acceptance), values-based actions, experiential avoidance, and cognitive/emotional fusion.
  Scoring: The AFQ-Y consists of 17 items. Scale range: Responses are rated on a Likert scale from 0 ("Not at all true") to 4 ("Very true").
  Interpretation: Higher scores indicate greater psychological inflexibility, which is considered a worse outcome.
Emotion Regulation Scale (DERS-36) | over the time period of one year of intervention, october to october
  This 36-item questionnaire measures various aspects of emotion regulation difficulties, including emotional awareness, clarity, acceptance, impulse control, goal-directed behavior, and access to regulation strategies.
  Scoring: Each item is rated from 1 ("Almost never") to 5 ("Almost always"). Scale range: Total scores range from 36 to 180. Interpretation: Higher scores indicate more severe difficulties in emotion regulation, reflecting a worse outcome.
Insomnia Severity Index (ISI) | over the time period of one year of intervention, october to october
  The ISI assesses the nature, severity, and impact of insomnia. It includes questions on sleep onset, sleep maintenance, early morning waking, satisfaction with sleep, and impact on daily functioning.
  Scoring: 7 items, each rated from 0 ("No problem") to 4 ("Very severe problem").
  Scale range: Total scores range from 0 to 28. Interpretation: Higher scores indicate more severe insomnia symptoms, a worse outcome.
Perceived Stress Scale - Youth Version (PSS-Y) | over the time period of one year of intervention, october to october
  This scale measures the degree to which situations in one's life are appraised as stressful, specifically for children and adolescents.
  Scoring: Items are typically rated on a 5-point Likert scale. Scale range: Depending on version, generally 0 to 40. Interpretation: Higher scores reflect greater perceived stress, a worse outcome.
WHO-5 Well-Being Index | over the time period of one year of intervention, october to october
  This short questionnaire assesses subjective psychological well-being over the past two weeks. It focuses on positive mood, vitality, and general interest.
  Scoring: 5 items, each scored from 0 ("At no time") to 5 ("All of the time"). Scale range: Raw scores range from 0 to 25, which are then multiplied by 4 to give a final score from 0 to 100.
  Interpretation: Higher scores indicate better well-being, a better outcome. Scores below 50 may indicate reduced well-being or risk of depression.
Accelerometer-Based Monitoring | over the time period of one year of intervention, october to october
  Physical activity is objectively measured over a 7-day period using a wrist-worn accelerometer. This device collects data on:
  Duration, frequency, and intensity of movement Data source: Integrated gyroscope and accelerometer sensors Interpretation: Data is analyzed in line with age-appropriate activity thresholds (e.g., moderate-to-vigorous physical activity levels)
Recall-Based Physical Activity Protocol | over the time period of one year of intervention, october to october
  Participants provide a structured recall of the types of physical activities they engaged in during different parts of the day over the same 7-day period. This qualitative input complements the accelerometer data and offers context about activity types and preferences.
International Physical Activity Questionnaire - Short Form (IPAQ-Short) | over the time period of one year of intervention, october to october
  This questionnaire assesses physical activity levels over the past 7 days, including walking, moderate activity, vigorous activity, and sitting time.
  Scoring: Time spent in each activity type is used to estimate energy expenditure in MET-minutes per week.
  Interpretation: Higher MET-minutes indicate higher physical activity, a better outcome.
Tanner Stages Self-Assessment Questionnaire | over the time period of one year of intervention, october to october
  To assess pubertal development, participants self-rate physical characteristics based on standardized illustrations and descriptions of secondary sexual characteristics (e.g., pubic hair, breast/genital development).
  Interpretation: Tanner stages range from Stage 1 (pre-pubertal) to Stage 5 (fully mature), allowing categorization into early, mid, or late pubertal status.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Roth, Phd, Principal Investigator — University of Basel, Department of Sport, Exercise and Health
Locations (1):
- Department of Sport, Exercise and Health, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No